CLINICAL TRIAL: NCT01754129
Title: Global REsponsE During iNFusIon of a gEl With LevoDopa/Carbidopa (GREENFIELD)
Brief Title: Global REsponsE During iNFusIon of a gEl With LevoDopa/Carbidopa
Acronym: GREENFIELD
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-895
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Parkinson's Disease
Keywords: Caregiver; Quality of Life; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Parkinson's disease: Participants with advanced levodopa-responsive Parkinson's disease and severe motor fluctuations and hyper-/dyskinesia who were prescribed and treated in accordance with the local levodopa/carbidopa intestinal gel product label

SUMMARY:
This multicenter, post marketing observational study (PMOS) was designed to evaluate the long-term effectiveness of levodopa/carbidopa intestinal gel (DUODOPA) on motor fluctuations (duration of OFF periods) in participants with advanced levodopa-responsive Parkinson's disease (PD) and severe motor fluctuations and hyper-/dyskinesia (involuntary movements). Secondary objectives of this study were to assess the participants' quality of life; to assess the long-term safety of DUODOPA; to assess disability, cognitive function, and non-professional caregiver burden; and to assess the economic and social impact of family caregiver assistance.

DETAILED DESCRIPTION:
Male or female participants ages 18 years of age who were already on DUODOPA treatment and had concluded the naso-intestinal phase were included in this study. DUODOPA was administered via a portable pump directly into the proximal small intestine via a percutaneous endoscopic transgastric jejunostomy (PEG-J) tube. There were 3 planned visits during the study: enrollment (Visit 1), 1 year (Visit 2), and 2 years (Visit 3).

ELIGIBILITY:
Inclusion Criteria:

* Participants already on treatment with DUODOPA (having already concluded the naso-intestinal treatment phase) according to the local DUODOPA product label and to routine clinical care for advanced PD patients
* Participants with available data on DUODOPA treatment, on previous PD conventional treatments and with at least one of the scales/questionnaires under study already collected on the participant's clinical chart
* Participant or legal representative has given written informed consent
* Non-professional caregiver (relative or familiar who give daily assistance to the patient) has given his/her written consent

Exclusion Criteria:

• History or presence of any condition that might interfere with the long-term continuation of the duodenal infusion of DUODOPA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants already on DUODOPA treatment in accordance with the local DUODOPA product label (treatment of advanced levodopa-responsive Parkinson's disease with severe motor fluctuations and hyper/dyskinesia when available combinations of PD medicinal products have not given satisfactory results) and according to specific reimbursement criteria were offered the opportunity to enroll in this study.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2012-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screened population: all participants who were screened for the study
Period: Overall Study
Arm/Group | Participants With Parkinson's Disease
Started | 148
Visit 1 (Enrollment Day) | 145
Visit 2 (Year 1) | 129
Visit 3 (Year 2) | 115
Completed | 115
Not Completed | 33
Not completed — Death | 13
Not completed — Duodopa discontinuation | 9
Not completed — Lost to Follow-up | 7
Not completed — Withdrew consent | 1
Not completed — Inclusion/exclusion criteria violation | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants from the screened population with all inclusion/exclusion criteria met
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (7.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 73
Time since Parkinson's disease diagnosis [Mean (Standard Deviation); unit: years] | 14.7 (6.46)
Time since onset of Parkinson's disease motor fluctuations [Mean (Standard Deviation); unit: years] | 5.9 (3.94)

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) IV (Complications of Therapy) Item 39 (Proportion of Waking Day Spent in "Off") Score: Mean Change From Baseline to the Last Available Follow up
Description: Section B of the UPDRS IV questionnaire consists of 4 individual items that assess the degree of clinical fluctuations. Item 39 is the percentage of "off" times (when PD symptoms are not adequately controlled by the drug) during the waking day. The Item 39 score ranges from 0 (None), 1 (1- 25% of the waking day), 2 (26 - 50% of the waking day), 3 (51 - 75% of the waking day), and 4 (76 - 100% of the waking day). The mean change from baseline was calculated as the score at the last available follow up visit minus the score at baseline/Visit 1. Negative change from baseline for "off" time indicates improvement.
Time Frame: Baseline/Visit 1 and Visit 2 (Year 1) or Visit 3 (Year 2)
Population: Evaluable population: participants with at least one post-baseline visit. Missing data at Visit 3 was replaced using Last Observation Carried Forward technique.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 135
units on a scale
  Change from baseline to Visit 3: number analyzed (Participants) | 130
  Change from baseline to Visit 3 | -0.97 [-1.15 to -0.79]
  Change from baseline to Visit 2: number analyzed (Participants) | 127
  Change from baseline to Visit 2 | -1.04 [-1.23 to -0.85]
Statistical Analysis 1: Comparison: Participants With Parkinson's Disease; Mean change from baseline to Visit 3; Test type: Other; p < 0.001, Paired t-test — Missing values were replaced using the Last Observation Carried Forward (LOCF) technique for data of questionnaires. Missing data at Visit 3 was replaced with the (non-missing) data recorded at Visit 2
Statistical Analysis 2: Comparison: Participants With Parkinson's Disease; Change from baseline to Visit 2; Test type: Other; p < 0.001, Paired t-test

2. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) IV (Complications of Therapy) Part A+B Score: Mean Change From Baseline to Visits 2 and 3
Description: The UPDRS is an Investigator-used rating tool to follow the course of Parkinson's disease. Scores for dyskinesias, early-morning dystonia, and clinical fluctuations ("off" times when PD symptoms are not adequately controlled by the drug) were assessed by the sum of the Part A+B items, questions 32-39. Questions 32-34 and 39 are measured on a 5-point scale (0-4), with 0 being no disease and 4 representing severe disease. Higher scores indicate a greater duration of dyskinesia (Q32), disability (Q33), and pain (Q34), and proportion of the waking day spent in "off" (Q39). Questions 35-38 are scored on a binary scale where 0= no and 1=yes, with higher scores indicating a higher incidence of early morning dystonia, and a higher degree of clinical fluctuations. The total score ranges from 0 (normal) to 20 (severe disease). Negative changes from baseline indicate improvement.
Time Frame: Baseline/Visit 1, Visit 2 (Year 1), and Visit 3 (Year 2)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 134
units on a scale
  Change from baseline to Visit 2: number analyzed (Participants) | 124
  Change from baseline to Visit 2 | -3.33 [-4.01 to -2.65]
  Change from baseline to Visit 3: number analyzed (Participants) | 128
  Change from baseline to Visit 3 | -3.08 [-3.72 to -2.43]

3. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale on Mentation, Behavior and Mood (UPDRS I) and Activities of Daily Living (UPDRS II) During On and Off Phases
Description: The UPDRS is an Investigator-used rating tool to follow the course of Parkinson's disease. The Part I Score is the sum of the answers to the 4 questions that comprise Part I, each of which are measured on a 5-point scale (0-4). The Part I score ranges from 0 to 16 and higher scores are associated with more disability. The Part II score is the sum of the answers to the 13 questions that comprise Part II, each of which are measured on a 5-point scale (0-4). The Part II score ranges from 0-52 and higher scores are associated with more disability. Scores for both "On" time (when PD symptoms are well-controlled by the drug) and "Off" time (when PD symptoms are not adequately controlled by the drug) are presented. Negative changes from baseline indicate improvement.
Time Frame: Baseline/Visit 1, Visit 2 (Year 1), and Visit 3 (Year 2)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 129
units on a scale
  UPDRS I "On" Change from baseline to Visit 2: number analyzed (Participants) | 126
  UPDRS I "On" Change from baseline to Visit 2 | -0.49 [-1.06 to 0.08]
  UPDRS I "On" Change from baseline to Visit 3 | -0.21 [-0.81 to 0.38]
  UPDRS I "Off" Change from baseline to Visit 2: number analyzed (Participants) | 81
  UPDRS I "Off" Change from baseline to Visit 2 | -0.83 [-1.68 to 0.01]
  UPDRS I "Off" Change from baseline to Visit 3: number analyzed (Participants) | 81
  UPDRS I "Off" Change from baseline to Visit 3 | -0.92 [-1.85 to 0.02]
  UPDRS II "On" Change from baseline to Visit 2: number analyzed (Participants) | 127
  UPDRS II "On" Change from baseline to Visit 2 | -2.42 [-3.98 to -0.86]
  UPDRS II "On" Change from baseline to Visit 3: number analyzed (Participants) | 128
  UPDRS II "On" Change from baseline to Visit 3 | -1.48 [-3.14 to 0.17]
  UPDRS II "Off" Change from baseline to Visit 2: number analyzed (Participants) | 86
  UPDRS II "Off" Change from baseline to Visit 2 | -3.79 [-5.66 to -1.92]
  UPDRS II "Off" Change from baseline to Visit 3: number analyzed (Participants) | 87
  UPDRS II "Off" Change from baseline to Visit 3 | -3.10 [-5.08 to -1.12]

4. Secondary Outcome: Change in Parkinson's Disease Quality of Life Questionnaire (PDQ-39) Scores
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in PD. These include: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. The total score is between 0 and 156, calculated as the total sum of the items, and higher scores are associated with more severe symptoms. Negative changes from baseline indicate improvement.
Time Frame: Baseline/Visit 1, Visit 2 (Year 1), and Visit 3 (Year 2)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 136
units on a scale
  Change from baseline to Visit 2: number analyzed (Participants) | 126
  Change from baseline to Visit 2 | -2.70 [-6.03 to 0.64]
  Change from baseline to Visit 3: number analyzed (Participants) | 131
  Change from baseline to Visit 3 | -0.09 [-3.28 to 3.10]

5. Secondary Outcome: Change in Parkinson's Disease Sleep Scale Version 2 (PDSS-2) Scores
Description: The Parkinson's Disease Sleep Scale version 2 (PDSS-2) is a self-administered 15-item questionnaire addressing sleep and nocturnal disturbances in PD, including sleep quality, difficulty falling and staying asleep, restlessness, pain, or muscle cramps in legs or arms, dreams or hallucinations, getting up at night to pass urine, immobility at night, painful posturing in the morning, tremor on waking, sleepiness upon waking, and snoring or breathing difficulties. Scores on each item range from 0 (never) to 4 (very frequent). The PDSS-2 total score ranges from 0 (no disturbance) to 60 (maximum nocturnal disturbance). Negative changes from baseline indicate improvement.
Time Frame: Baseline/Visit 1, Visit 2 (Year 1), and Visit 3 (Year 2)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 135
units on a scale
  Change from baseline to Visit 2: number analyzed (Participants) | 125
  Change from baseline to Visit 2 | -1.19 [-2.59 to 0.20]
  Change from baseline to Visit 3: number analyzed (Participants) | 131
  Change from baseline to Visit 3 | -0.95 [-2.61 to 0.70]

6. Secondary Outcome: Change in Gait and Falls Questionnaire (GFQ) Scores
Description: The Gait and Falls questionnaire (GFQ) is a self-administered 16-item questionnaire addressing gait in daily living, the frequency and severity of freezing of gait, the frequency of festinating gait and its relation to falls, and the frequency and severity of falls. Scores on each item range from 0 (no symptoms) to 4 (severe symptoms). The GFQ total score ranges from 0 (normal function) to 64 (severely impaired function). Negative changes from baseline indicate improvement.
Time Frame: Baseline/Visit 1, Visit 2 (Year 1), and Visit 3 (Year 2)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 133
units on a scale
  Change from baseline to Visit 2 | -1.70 [-3.72 to 0.33]
  Change from baseline to Visit 3 | -0.81 [-3.03 to 1.40]

7. Secondary Outcome: Change in Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS) Scores
Description: The Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale is a 28-item survey used to assess the frequency and severity of behaviors including gambling, sexual behavior, buying, eating, performing tasks or hobbies, repeating simple activities, and PD medication use. Scores on each item range from 0 (never) to 4 (very often). The QUIP-RS total score ranges from 0 (normal function) to 112 (severely impaired function). Negative changes from baseline indicate improvement.
Time Frame: Baseline/Visit 1, Visit 2 (Year 1), and Visit 3 (Year 2)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 136
units on a scale
  Change from baseline to Visit 2 | -1.62 [-3.21 to -0.03]
  Change from baseline to Visit 3 | -2.02 [-3.76 to -0.27]

8. Secondary Outcome: Economic and Social Impact of Family-provided Healthcare
Description: Family caregivers were surveyed regarding the participant's need for home health care for Parkinson's Disease; the amount of time dedicated to care each week; the need of a family caregiver to reduce or change their normal work hours in order to provide care; the number of working days per month spent performing caregiver responsibilities; the number of hours of professional assistance per week needed; and the hourly costs of professional assistance incurred per week.
Time Frame: Baseline/Visit 1, Visit 2 (Year 1), and Visit 3 (Year 2)
Population: Evaluable population: participants with at least one post-baseline visit
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Participants With Parkinson's Disease- Visit 1; Participants With Parkinson's Disease- Visit 2; Partcipants With Parkinson's Disease- Visit 3: Participants with advanced levodopa-responsive Parkinson's disease and severe motor fluctuations and hyper-/dyskinesia who were prescribed and treated in accordance with the local levodopa/carbidopa intestinal gel product label
Arm/Group | Participants With Parkinson's Disease- Visit 1 | Participants With Parkinson's Disease- Visit 2 | Partcipants With Parkinson's Disease- Visit 3
Number analyzed (Participants) | 137 | 129 | 115
hours
  Hours/week of care provided by family caregiver | 51 (54) | 52.4 (54) | 53 (56)
  Work hours/week lost by family caregiver | 23.6 (23) | 21.3 (26.1) | 21.7 (22.5)
  Hours/week of professional assistance | 44.1 (54.7) | 32 (41.4) | 32 (42)

9. Secondary Outcome: Change in Relative Stress Scale (RSS) Scores
Description: The Relative Stress Scale is a 15-item questionnaire completed by family caregivers to assess personal distress, life upset, and negative feelings regarding caring for a family member with PD. Scores on each item range from 1 (not at all) to 5 (to a high degree). The RSS total score ranges from 15 (low stress) to 75 (severe stress). Negative changes from baseline indicate improvement.
Time Frame: Baseline/Visit 1, Visit 2 (Year 1), and Visit 3 (Year 2)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 133
units on a scale
  Change from baseline to Visit 2: number analyzed (Participants) | 123
  Change from baseline to Visit 2 | -0.20 [-1.56 to 1.17]
  Change from baseline to Visit 3: number analyzed (Participants) | 126
  Change from baseline to Visit 3 | 0.09 [-1.58 to 1.76]

10. Secondary Outcome: Concomitant Diseases and Medications
Description: Concomitant diseases were coded using the MedDRA dictionary (version 15.1). Concomitant diseases present in ≥ 5% of participants started before or at Visit 1 and stopped after Visit 1 or ongoing or started after Visit 1 are presented. Non-PD medications in ≥ 5% of participants maintained with a start date previous to the date of Visit 1 and a stop date after date of Visit 1 or ongoing are listed.
Time Frame: Baseline/Visit 1, Visit 2 (Year 1), and Visit 3 (Year 2)
Population: All enrolled participants from the screened population with all inclusion/exclusion criteria met
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 145
Participants
  Hypertension | 34
  Depression | 22
  Carpal tunnel syndrome | 9
  Diabetes mellitus | 11
  Hypothyroidism | 8
  Clozapine | 11
  Quetiapine fumarate | 10
  Clonazepam | 10
  Acetylsalicylic acid | 12
  Folic acid | 8

11. Secondary Outcome: Change in Global Effectiveness on Motor Symptoms as Compared to Baseline
Description: Motor symptoms were rated by neurologists using three categories: improvement, no change, or worsening as compared to symptoms present at baseline.
Time Frame: Baseline/Visit 1, Visit 2 (Year 1), and Visit 3 (Year 2)
Population: Evaluable population: participants with at least one post-baseline visit
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Parkinson's Disease- Visit 1 | Participants With Parkinson's Disease- Visit 2 | Partcipants With Parkinson's Disease- Visit 3
Number analyzed (Participants) | 137 | 129 | 115
Participants
  Worsening | 3 | 7 | 5
  No change | 2 | 13 | 22
  Improvement | 132 | 107 | 87
  Missing | 0 | 2 | 1

12. Secondary Outcome: Participant Self-assessment Scale of DUODOPA Therapy
Description: Participants were asked to rate DUODOPA therapy on a scale from 0 to 10 (0-2 worse, 3-5, unsatisfactory, 6-8 satisfactory, 9-10, very good).
Time Frame: Baseline/Visit 1, Visit 2 (Year 1), and Visit 3 (Year 2)
Population: Evaluable population: participants with at least one post-baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Parkinson's Disease
Number analyzed (Participants) | 137
units on a scale
  Visit 1 | 7.1 (1.60)
  Visit 2: number analyzed (Participants) | 125
  Visit 2 | 7.1 (1.37)
  Visit 3: number analyzed (Participants) | 113
  Visit 3 | 7.0 (1.26)

13. Secondary Outcome: DUODOPA Total Daily Infusion Dosage
Description: The total daily DUODOPA infusion dosage was documented at study visits starting at the baseline visit. One mL of DUODOPA contains 20 mg levodopa and 5 mg carbidopa monohydrate.
Time Frame: Baseline, Visit 1, Visit 2, (Year 1) and Visit 3 (Year 2)
Population: Evaluable population: participants with at least one post-baseline visit
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Participants With Parkinson's Disease- Baseline; Participants With Parkinson's Disease- Visit 1; Partcipants With Parkinson's Disease- Visit 2; Partcipants With Parkinson's Disease- Visit 3: Participants with advanced levodopa-responsive Parkinson's disease and severe motor fluctuations and hyper-/dyskinesia who were prescribed and treated in accordance with the local levodopa/carbidopa intestinal gel product label
Arm/Group | Participants With Parkinson's Disease- Baseline | Participants With Parkinson's Disease- Visit 1 | Partcipants With Parkinson's Disease- Visit 2 | Partcipants With Parkinson's Disease- Visit 3
Number analyzed (Participants) | 133 | 143 | 124 | 113
mL | 56.37 (20.14) | 56.61 (20.98) | 58.91 (17.61) | 58.8 (17.67)

ADVERSE EVENTS:
Time Frame: Treatment emergent serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 108 weeks).
Description: Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Participants With Parkinson's Disease
Serious Adverse Events (participants affected / at risk) | 40/145
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Parkinson's Disease (N=145)
Pneumonia (Infections and infestations) | 4
Peritonitis (Infections and infestations) | 2
Administration site infection (Infections and infestations) | 1
Stoma site infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 3
Wrong technique in drug usage process (Injury, poisoning and procedural complications) | 2
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Parkinson's disease (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Cerebral haematoma (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hyperkinesia (Nervous system disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Cardiac arrest (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Death (General disorders) | 2
Device occlusion (General disorders) | 1
Medical device complication (General disorders) | 1
Pyrexia (General disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Agitation (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.